CLINICAL TRIAL: NCT05969054
Title: A Clinical Study Exploring Lacosamide and Levetiracetam in Improving Cognitive in Patients With Alzheimer's Disease and Epilepsy
Brief Title: Improvement Effect of Lacosamide and Levetiracetam on Cognitive in Alzheimer's Disease Patients With Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Feng, MD, PhD, Associate Professor Vice Direct of Neurology Teaching and Research Office, Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202306123
Record Dates: First submitted 2023-07-12; First posted 2023-08-01 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer Disease 3; Epilepsy
Keywords: Alzheimer Disease; Epilepsy; lacosamide; levetiracetam
MeSH Terms: conditions — Alzheimer disease, familial, type 3; Epilepsy; Alzheimer Disease | interventions — Lacosamide; Levetiracetam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: lacosamide (Experimental): Subjects who were randomly divided into group A took lacosamide for 6 months during treatment (initial dose was 50mg bid, maintained for one week and then increased to 100mg bid and maintained at this dose)
  Interventions: Drug: Lacosamide 100 mg
- Group B: levetiracetam (Experimental): Subjects randomly divided into group B took levetiracetam for 6 months during treatment (initial dose was 250mg bid, maintained for one week and then increased to 500mg bid and maintained at this dose).
  Interventions: Drug: Levetiracetam 250mg

INTERVENTIONS:
Drug: Lacosamide 100 mg — Subjects who were randomly divided into group A took lacosamide for 6 months during treatment (initial dose was 50mg bid, maintained for one week and then increased to 100mg bid and maintained at this dose)
  Arms: Group A: lacosamide
Drug: Levetiracetam 250mg — Subjects randomly divided into group B took levetiracetam for 6 months during treatment (initial dose was 250mg bid, maintained for one week and then increased to 500mg bid and maintained at this dose).
  Arms: Group B: levetiracetam

SUMMARY:
Participants will perform Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Clinical Dementia Rating (CDR), Alzheimer's disease assessment scale-cognitive section (ADAS-Cog), Hamilton Anxiety Scale (HAMA) and Hamilton Depression Rating Scale (HAMD) evaluation. The patients will be randomly divided into two groups, treated with lacosamide and levetiracetam respectively, and maintained for 6 months.

Researchers will compare the lacosamide group with the levetiracetam group to see if the improvement of cognitive function in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as Alzheimer's disease and treated with cholinesterase inhibitors;
* New seizures or subclinical epileptic discharges;
* Mini-Mental State Examination score ≥ 18 points, and/or Clinical Dementia Rating (CDR) score < 2 points;
* Sign the informed consent form.

Exclusion Criteria:

* Suffering from syncope, transient ischemic attack, hysteria attack, migraine and other transient brain dysfunction;
* Serious medical disease (especially atrioventricular block) or mental illness;
* There are structural abnormalities related to epilepsy in other brain regions of imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | At the time of enrollment
  The minimum value is 0, the maximum value is 30, the higher scores means a better cognition.
Mini-Mental State Examination (MMSE) | 1 month after enrollment
  The minimum value is 0, the maximum value is 30, the higher scores means a better cognition.
Mini-Mental State Examination (MMSE) | 3 months after enrollment
  The minimum value is 0, the maximum value is 30, the higher scores means a better cognition.
Mini-Mental State Examination (MMSE) | 6 months after enrollment
  The minimum value is 0, the maximum value is 30, the higher scores means a better cognition.
Montreal Cognitive Assessment (MoCA) | At the time of enrollment
  The minimum value is 0, the maximum value is 30, the higher score means a better cognition.
Montreal Cognitive Assessment (MoCA) | 1 month after enrollment
  The minimum value is 0, the maximum value is 30, the higher score means a better cognition.
Montreal Cognitive Assessment (MoCA) | 3 months after enrollment
  The minimum value is 0, the maximum value is 30, the higher score means a better cognition.
Montreal Cognitive Assessment (MoCA) | 6 months after enrollment
  The minimum value is 0, the maximum value is 30, the higher score means a better cognition.
Clinical Dementia Rating (CDR) | At the time of enrollment
  The minimum value is 0, the maximum value is 3, the higher scores means a great likelihood of dementia.
Clinical Dementia Rating (CDR) | 1 month after enrollment
  The minimum value is 0, the maximum value is 3, the higher scores means a great likelihood of dementia.
Clinical Dementia Rating (CDR) | 3 months after enrollment
  The minimum value is 0, the maximum value is 3, the higher scores means a great likelihood of dementia.
Clinical Dementia Rating (CDR) | 6 months after enrollment
  The minimum value is 0, the maximum value is 3, the higher scores means a great likelihood of dementia.
Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) scale | At the time of enrollment
  The minimum value is 0, the maximum value is 75, the higher scores means a great likelihood of dementia
Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) scale | 1 month after enrollment
  The minimum value is 0, the maximum value is 75, the higher scores means a great likelihood of dementia
Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) scale | 3 months after enrollment
  The minimum value is 0, the maximum value is 75, the higher scores means a great likelihood of dementia
Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog) scale | 6 months after enrollment
  The minimum value is 0, the maximum value is 75, the higher scores means a great likelihood of dementia
Hamilton Anxiety Scale (HAMA) | At the time of enrollment
  The minimum value is 0, the maximum value is 56, the higher scores means a great likelihood of anxiety
Hamilton Anxiety Scale (HAMA) | 1 month after enrollment
  The minimum value is 0, the maximum value is 56, the higher scores means a great likelihood of anxiety
Hamilton Anxiety Scale (HAMA) | 3 months after enrollment
  The minimum value is 0, the maximum value is 56, the higher scores means a great likelihood of anxiety
Hamilton Anxiety Scale (HAMA) | 6 months after enrollment
  The minimum value is 0, the maximum value is 56, the higher scores means a great likelihood of anxiety
Hamilton Depression Scale (HAMD) | At the time of enrollment
  The minimum value is 0, the maximum value is 77, the higher scores means a great likelihood of depression
Hamilton Depression Scale (HAMD) | 1 month after enrollment
  The minimum value is 0, the maximum value is 77, the higher scores means a great likelihood of depression
Hamilton Depression Scale (HAMD) | 3 months after enrollment
  The minimum value is 0, the maximum value is 77, the higher scores means a great likelihood of depression
Hamilton Depression Scale (HAMD) | 6 months after enrollment
  The minimum value is 0, the maximum value is 77, the higher scores means a great likelihood of depression

SECONDARY OUTCOMES:
Seizure frequency | At the time of enrollment
  Record seizure frequency
Seizure frequency | 1 month after enrollment
  Record seizure frequency
Seizure frequency | 3 months after enrollment
  Record seizure frequency
Seizure frequency | 6 months after enrollment
  Record seizure frequency
EEG discharge | At the time of enrollment
  Record interictal epileptic discharge under the 24-hour VEEG
EEG discharge | 1 month after enrollment
  Record interictal epileptic discharge under the 24-hour VEEG
EEG discharge | 3 months after enrollment
  Record interictal epileptic discharge under the 24-hour VEEG
EEG discharge | 6 months after enrollment
  Record interictal epileptic discharge under the 24-hour VEEG

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China